CLINICAL TRIAL: NCT06063564
Title: Adapting and Testing a Novel Digital Health Tool (PREVENT) to Improve Health Behavior Counseling and Cardiovascular Health in Rural Primary Care Clinics
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 202307156
Record Dates: First submitted 2023-09-20; First posted 2023-10-02 (Actual); Last update posted 2025-10-16 (Actual); Status verified 2025-10

CONDITIONS: Obesity; Cardiovascular Diseases
MeSH Terms: conditions — Obesity; Cardiovascular Diseases

STUDY DESIGN:
Intervention Model Description: Clinic randomized trial
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Wait-List Control (Active Comparator): Complete questionnaires at baseline (administered electronically or by mail). Follow-up measures will be administered immediately following their clinic visit and at 6-months after the clinic visit electronically and by mail. A PREVENT action plan (behavior change prescription, community resources, and education) will be provided to the patient via email after the completion of the follow-up measurement.
  Interventions: Behavioral: Wait-list Control
- PREVENT Intervention (Experimental): Complete questionnaires at baseline (administered electronically or by mail). Follow-up measures will be administered immediately following the clinic visit, and monthly for 6-months after the clinic visit electronically and by mail
  At the clinic visit, the provider will use the PREVENT tool to discuss CVH risk. A community health worker (CHW) will deliver a tailored behavioral change plan inclusive of patient-centered community resources. The CHW will provide ongoing support with goals and social needs for 6-months.
  Interventions: Behavioral: PREVENT

INTERVENTIONS:
Behavioral: PREVENT — PREVENT is a novel Health Information Technology tool designed to promote physical activity and healthy food intake among overweight/obese patients at the point of care. PREVENT automates the delivery of personalized, evidence-based behavior change recommendations and provides an interactive map of community resources to help providers link patients to resources in their community.
  Arms: PREVENT Intervention
Behavioral: Wait-list Control — Will receive routine clinical care. After completion of follow-up measures, control participants will receive a behavior change prescription via the PREVENT tool.
  Arms: Wait-List Control

SUMMARY:
The focus on this application is low-income, rural patients, since cardiovascular disease (CVD) prevalence is 40% higher among rural than urban residents. Health behavior counseling and follow-up care are required for patients with an elevated body mass index who have increased risk for CVD. Counseling is most effective when developed with, and tailored to, the patient and offered with resources that support healthy food intake and physical activity. Resource referral and follow-up is particularly important in rural low income residents who often have more severe social needs that impede healthy behaviors. The proposed research will leverage the candidate's digital health tool (PREVENT) for healthcare teams to use within the clinic visit. PREVENT visually displays patient-reported and electronic health record (EHR) data to facilitate counseling and deliver tailored physical activity and healthy food intake goals and resources. PREVENT may improve the quality of required care and promote cardiovascular health equity. This research will: 1) collaborate with rural and clinic partners to modify and integrate the PREVENT tool for low-income, rural patients with obesity (Aim 1); and 2) conduct a pilot pragmatic clinical trial of PREVENT to optimize feasibility, acceptability, appropriateness, and potential health equity impact.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-64 years at baseline
* a BMI ≥ 30
* Receiving care from the Missouri Highlands.
* Ability to understand and willingness to sign an IRB approved written informed consent document (or that of legally authorized representative, if applicable).

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-08-20 (Actual); Primary Completion 2028-01-31 (Estimated); Study Completion 2028-01-31 (Estimated)

PRIMARY OUTCOMES:
Patients' satisfaction of PREVENT tool: survey | 6-months
  A survey (6-questions) will assess patient's satisfaction with the PREVENT tool. Questions are asked on a 5-point Likert scale (range: 6-30) with a higher score indicating greater satisfaction.
Provider's satisfaction of PREVENT tool: survey | Up to 12 weeks post-study
  A survey (31-questions) will assess provider's acceptability and satisfaction with five aspects of health information technology: content, accuracy, format, ease of use and timeliness. Questions are asked on a 5-point Likert scale (range: 31-155) with a higher score indicating greater satisfaction.
Fidelity of PREVENT tool implementation | 0-6 months
  Fidelity will be measured using direct observation of patient-provider interactions while using the PREVENT tool. A direct observation checklist will be used by the observer to determine the number of interactions with the PREVENT tool that were implemented as intended.

SECONDARY OUTCOMES:
Change in provider confidence: survey | At baseline, and 6-months
  Provider confidence in discussing CVH and health behaviors with overweight and obese patients will be assessed using a survey (4-questions). Questions are asked on 5-point Likert scale (range: 4-20) with a higher score indicating greater confidence.
Quality of health behavior counseling | Immediately following clinic visit
  Patient perceptions of the clinical interaction in which CVH and health behaviors will be assessed using a survey (10- questions). Questions are asked as yes/no/I don't' know. Quality counseling will be defined as patient reported yes to their care team: 1) talking to them about healthy food intake; 2) talking to them about physical activity 3) delivering goals and 4) delivering resources.
Change in patient's motivation | At baseline, 3 months and 6-months
  A survey (15-question) administered to patients will assess motivation and self-efficacy for behavior change. Questions are asked using a 5-point Likert scale (range: 15-75) with a higher score indicating greater motivation.
Change in food intake behaviors | At baseline, 3 months and 6-months
  Patient-reported food intake behaviors (fruit and vegetable intake, whole grains, sugar-sweetened beverages and snacking behaviors) are collected using a brief Health Behavior & Attitudes Survey.
Change in minutes of moderate to vigorous physical activity | At baseline, 3 months and 6-months
  Patient-reported physical activity (minutes of moderate and vigorous activity per week) are collected using a survey (4-questions). Patients report the average number of minutes of moderate and vigorous activity they do per week.
Change in body mass index (BMI) | At baseline, and 6-months
  Collected from patient's medical record.
Change on patient's average systolic and diastolic blood pressure | At baseline, and 6-months
  Collected from patient's medical record.
Change in patient's cholesterol | At baseline, and 6-months
  Collected from patient's medical record.
Change in patient's blood glucose | At baseline, and 6-months
  Collected from patient's medical record.

CONTACTS AND LOCATIONS:
Locations (1):
- Washington University in St. Louis, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No